CLINICAL TRIAL: NCT03568877
Title: Anti-obesity Effects of Metabolaid® With AMPK-activating Capacity in Overweight Subjects: A Randomized Controlled Trial
Brief Title: Effect of Metabolaid® on AMPK Activation for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Monteloeder SL (Unknown)
Responsible Party: Principal Investigator, María Herranz-Lopez, Assistant Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UniversidadMHE_Met AMPK
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator): 2 capsules per day, each with 400 mg Cellulose microcrystalline, for 8 weeks
  Interventions: Dietary Supplement: Placebo
- Dietetic Supplement Group (Experimental): 2 Capsules per day of Metabolaid® (each capsule contains 250 mg Metabolaid®, 150 mg cellulose microcrystalline), for 8 weeks
  Interventions: Dietary Supplement: Metabolaid®

INTERVENTIONS:
Dietary Supplement: Metabolaid® — 500 mg per day, in fasting conditions.
  Arms: Dietetic Supplement Group
Dietary Supplement: Placebo — 500 mg per day, in fasting conditions.
  Arms: Placebo Control

SUMMARY:
The objective of this study was to establish a formulation, containing both Hibiscus sabdariffa L. (HS) and Lippia citriodora L. (LC) extracts (Metabolaid®) that had significant capacity to activate the AMPK-enzyme and to reduce triglyceride accumulation in the hypertrophied adipocyte model. Then, we assessed the efficacy of this combination in light-to-moderate-overweight subjects under risk of developing metabolic syndrome.

DETAILED DESCRIPTION:
AMP-activated protein kinase (AMPK) has been postulated as a molecular target in the amelioration of obesity-related diseases, where most therapeutic approaches have failed. Plant-polyphenols have shown the capacity to ameliorate obesity-induced metabolic disturbances. A combination of polyphenols (LC-HS) derived from Hibiscus sabdariffa L. (HS) and Lippia citriodora L. (LC) (lemon verbena) (Metabolaid®) was assessed for triglyceride accumulation and AMPK activation in the hypertrophied adipocyte model 3T3-L1. A dietary supplement containing 500 mg of LC-HS was evaluated in a double blind, placebo-controlled and randomized trial in 56 overweight subjects for two months. Anthropometric and circulating biochemical parameters were determined.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a body mass index (BMI) from 24 to 34 kg/m2

Exclusion Criteria:

* total cholesterol lower than 200 mg/dL.
* use of prescription medication for cholesterol or hypertension.
* presence of any obesity-related pathology.
* hormone replacement therapy.
* consumption of antioxidant supplements/drugs.
* alcohol addiction.
* women who were pregnant or lactating.

Ages: 36 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in body Weight, using a weight scale | At the beginning, four weeks and end of the intervention, total eight weeks.
  In Kg

SECONDARY OUTCOMES:
Height, using measuring tape | At the beginning, four weeks and eight weeks
  In cm
BMI, calculated based on Weight and Height | At the beginning, four weeks and eight weeks
  in kg/m^2
Waist Circumference, using a measuring tape | At the beginning, four weeks and eight weeks
  in kg/m^2
Glucose | At the beginning, four weeks and eight weeks
  Blood Sampling in Fasting conditions, in mg/dl
Tryglicerides | At the beginning, four weeks and eight weeks
  Blood Sampling in Fasting conditions, in mg/dl
LDL Cholesterol | At the beginning, four weeks and eight weeks
  Blood Sampling in Fasting conditions, in mg/dl
HDL Cholesterol | At the beginning, four weeks and eight weeks
  Blood Sampling in Fasting conditions, in mg/dl
Total Cholesterol | At the beginning, four weeks and eight weeks
  Blood Sampling in Fasting conditions, in mg/dl
Blood Pressure | At the beginning, four weeks and eight weeks
  Single Blood Pressure measurements, using the Omron M6 Comfort device
Heart rate | At the beginning, four weeks and eight weeks
  Single Blood Pressure measurements, using the Omron M6 Comfort device

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernandez de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No